CLINICAL TRIAL: NCT00638443
Title: Lumbar Stenosis Outcomes Research (LUSTOR)- A Randomized, Double-blind, Cross-over Trial of Pregabalin vs. Diphenhydramine in Patients With Lumbar Spinal Stenosis and Neuropathic Low Back Pain
Brief Title: Lumbar Stenosis Outcomes Research (LUSTOR)
Acronym: LUSTOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, John Markman, Director, Translational Pain Research, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 16697; IIR#GA00818X (Other: Sponsor ID)
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-05

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Neurogenic claudication, lumbar spinal stenosis, treadmill testing
MeSH Terms: conditions — Spinal Stenosis | interventions — Pregabalin; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin then Diphenhydramine (Other): Pregabalin started at 75mg twice daily for 3 days; pregabalin increased to 150mg twice daily for 7 days; pregabalin reduced to 75mg twice daily for 3 days; no drug for 7 days; diphenhydramine started at 6.25mg twice daily for 3 days; diphenhydramine increased to 12.5mg twice daily for 7 days; diphenhydramine reduced to 6.25mg twice daily for 3 days.
  Interventions: Drug: Pregabalin; Drug: Diphenhydramine
- Diphenhydramine then Pregabalin (Other): diphenhydramine started at 6.25mg twice daily for 3 days; diphenhydramine increased to 12.5mg twice daily for 7 days; diphenhydramine reduced to 6.25mg twice daily for 3 days; no drug for 7 days; pregabalin started at 75mg twice daily for 3 days; pregabalin increased to 150mg twice daily for 7 days; pregabalin reduced to 75mg twice daily for 3 days.
  Interventions: Drug: Pregabalin; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Pregabalin — Pregabalin started at 75mg twice daily for 3 days; pregabalin increased to 150mg twice daily for 7 days; pregabalin reduced to 75mg twice daily for 3 days.
  Other Names: Lyrica
Drug: Diphenhydramine — diphenhydramine started at 6.25mg twice daily for 3 days; diphenhydramine increased to 12.5mg twice daily for 7 days; diphenhydramine reduced to 6.25mg twice daily for 3 days.
  Other Names: Benedryl

SUMMARY:
The primary objective of the proposed pilot study is to determine the efficacy of pregabalin in prolonging the time to onset of pain and reducing the severity of pain associated with walking in patients with neurogenic claudication. Neurogenic claudication is defined as movement induced leg pain, numbness, heaviness, or vague discomfort in part or all of one or both legs provoked with walking and standing and relieved by sitting, squatting, or forward flexion posturing. The secondary objective is to examine the functional benefit of pregabalin with respect to improvement in duration and distance of walking.

DETAILED DESCRIPTION:
Subjects were randomized into one of two treatment sequences: pregabalin/active placebo or active placebo/pregabalin. Each arm lasted 10 days, with a washout period of 10 days between treatments. Pregabalin was administered as a standardized two step titration, starting at 75mg twice daily up to a maximum daily dose of 150mg twice daily; and likewise, diphenhydramine (active placebo) was administered starting at 6.25mg twice daily up to a maximum daily dose of 12.5mg twice daily. The primary endpoint was time to first symptoms of moderate intensity (NRS ≥ 4/10) during treadmill ambulation. Ambulation assessment was performed during the screening visit, and on day 10 of each period to evaluate pain intensity associated with walking as well as distance covered by the patients. Quantitative assessment of ambulation was conducted on a treadmill at 0° ramp incline at 1.2 miles per hour (mph). Measurement of self-reported symptom severity using the NRS at baseline, and every 30 seconds for a maximum of 15 minutes was recorded. The following information was also recorded: time to first symptoms, total ambulation time. The examination was stopped after 15 minutes or at the onset of severe symptoms. Severe symptoms were defined as the level of discomfort that would make patients stop walking in usual life situations. No one was encouraged or prompted to continue walking beyond this point. Patients were instructed to walk with an upright posture. They were not permitted to lean forward or hold onto the handrails during the examination. Secondary outcome measures included area under the curve of present pain intensity with ambulation at each specified time point, final pain intensity with walking, walking tolerance, time to return to baseline pain level after ambulation, as well as the results of a series of pain related questionnaires including: Visual Analog Scale (VAS), Patient Global Assessment (PGA), NRS, Roland Morris Disability Questionnaire (RMDQ), modified Brief Pain Inventory short form (mBPI-sf), Oswestry Disability Index (ODI), and Swiss Spinal Stenosis (SSS).

ELIGIBILITY:
Inclusion Criteria:

* Patients must present with clinical symptoms of neurogenic claudication (neurogenic claudication is defined as movement induced leg pain, numbness, heaviness, or vague discomfort in part or all of one or both legs provoked with walking and standing and relieved by sitting, squatting, or forward flexion posturing) and endorse limitation of walking tolerance due to these symptoms
* Numeric Rating Scale (NRS) for pain greater than or equal to 6 in response to the following questions: "Circle one number (from 0=no pain to 10=worst pain)-How would you rate the worst leg and lower back pain you experienced during walking last week?"
* Patients must have confirmatory imaging by MRI or CT scan demonstrating at least one level of lumbar spinal stenosis within 1 year
* Duration of symptoms > 3 months
* Age > 50 years; male or female

Exclusion Criteria:

* Past or present existence of movement disorder, e.g., Parkinsonism,or a neurologic disease that might affect the ability to ambulate (e.g., signs/symptoms of cauda equina compression)
* Cognitive impairment preventing full understanding or participation in the study
* Peripheral vascular disease
* Moderate to severe arthritis of the knee or hip that might severely compromise ambulation
* Past or present lower extremity peripheral vascular disease
* Serious concomitant medical illness (e.g., heart disease) that might impair ambulation assessment
* Previous lumbar surgery for spinal stenosis (laminectomy with or without fusion) within the past 2 years
* Prior treatment with study drug for neurogenic claudication
* Severe psychiatric disorder
* Mean time to severe symptoms > 15 minutes.
* Epidural steroid treatment within the last three months
* Ongoing treatment with gabapentin
* Hypersensitivity or allergic reaction to diphenhydramine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Markman, M.D, Principal Investigator — University of Rochester
Locations (1):
- 2180 South Clinton Avenue, Rochester, New York, United States

REFERENCES:
- [Background] Simon LS, Evans C, Katz N, Bombardier C, West C, Robbins J, Copley-Merriman C, Markman J, Coombs JH. Preliminary development of a responder index for chronic low back pain. J Rheumatol. 2007 Jun;34(6):1386-91. PMID 17552065
- [Background] Markman JD, Dworkin RH. Ion channel targets and treatment efficacy in neuropathic pain. J Pain. 2006 Jan;7(1 Suppl 1):S38-47. doi: 10.1016/j.jpain.2005.09.008. PMID 16427000
- [Background] Deen HG Jr, Zimmerman RS, Lyons MK, McPhee MC, Verheijde JL, Lemens SM. Test-retest reproducibility of the exercise treadmill examination in lumbar spinal stenosis. Mayo Clin Proc. 2000 Oct;75(10):1002-7. doi: 10.4065/75.10.1002. PMID 11040847
- [Background] Deen HG, Zimmerman RS, Lyons MK, McPhee MC, Verheijde JL, Lemens SM. Use of the exercise treadmill to measure baseline functional status and surgical outcome in patients with severe lumbar spinal stenosis. Spine (Phila Pa 1976). 1998 Jan 15;23(2):244-8. doi: 10.1097/00007632-199801150-00019. PMID 9474733
- [Background] Stucki G, Daltroy L, Liang MH, Lipson SJ, Fossel AH, Katz JN. Measurement properties of a self-administered outcome measure in lumbar spinal stenosis. Spine (Phila Pa 1976). 1996 Apr 1;21(7):796-803. doi: 10.1097/00007632-199604010-00004. PMID 8779009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Neuromedicine Pain Treatment Center between May 2008 and February 2010
Pre-assignment Details: 33 participants recruited; 4 excluded (did not meet inclusion criteria based on evoked pain being less than moderate intensity during treadmill ambulation).
Groups:
- Pregabalin First, Diphenhydramine Second: Pregabalin started at 75mg twice daily for 3 days; pregabalin increased to 150mg twice daily for 7 days; pregabalin reduced to 75mg twice daily for 3 days; washout 7 days; Diphenhydramine started at 6.25mg twice daily for 3 days; diphenhydramine increased to 12.5mg twice daily for 7 days; diphenhydramine reduced to 6.25mg twice daily for 3 days
- Diphenhydramine First, Pregabalin Second: Diphenhydramine started at 6.25mg twice daily for 3 days; diphenhydramine increased to 12.5mg twice daily for 7 days; diphenhydramine reduced to 6.25mg twice daily for 3 days; washout 7 days; Pregabalin started at 75mg twice daily for 3 days; pregabalin increased to 150mg twice daily for 7 days; pregabalin reduced to 75mg twice daily for 3 days.
Period: First Intervention
Arm/Group | Pregabalin First, Diphenhydramine Second | Diphenhydramine First, Pregabalin Second
Started | 14 | 15
Completed | 12 | 14
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1
Period: Washout
Arm/Group | Pregabalin First, Diphenhydramine Second | Diphenhydramine First, Pregabalin Second
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Pregabalin First, Diphenhydramine Second | Diphenhydramine First, Pregabalin Second
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Pregabalin started at 75mg twice daily for 3 days; pregabalin increased to 150mg twice daily for 7 days; pregabalin reduced to 75mg twice daily for 3 days
  Diphenhydramine started at 6.25mg twice daily for 3 days; diphenhydramine increased to 12.5mg twice daily for 7 days; diphenhydramine reduced to 6.25mg twice daily for 3 days
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.76 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Time to First Symptoms of Moderate Pain
Description: Using the Numeric Rating Scale (NRS) (0=no pain, 10=worst pain imaginable)the time to first symptoms (Tfirst) with a NRS score greater than or equal to 4 (moderate pain level), with treadmill ambulation was measured.
Time Frame: 10 days
Population: The analyses included all enrolled randomized subjects according to the inclusion and exclusion criteria except for the three who withdrew from the trial prior to the completion of the study. One dropped out of the study due to an adverse event (dizziness).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
minutes | 2.52 (2.83) | 3.06 (3.11)

2. Secondary Outcome: Final Pain as Measured by NRS
Description: Subjects were instructed to walk on the treadmill and to tell the research coordinator to stop testing when they reached the point at which they typically would need to stop and sit down, or until 15 minutes had elapsed. At defined intervals subjects were asked what their pain level was according to the NRS. When the subject reached their maximum distance, they were asked their NRS score. This was recorded as final pain intensity. Using the Numeric Rating Scale (NRS) (0=no pain, 10=worst pain imaginable)the time to first symptoms (Tfirst) with a NRS score greater than or equal to 4 (moderate pain level), with treadmill ambulation was measured.
Time Frame: 10 days
Population: Outcome measures were obtained for all subjects as described in the Analysis Population Description of the primary outcome above.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale | 1.82 (.35) | 1.53 (.35)

3. Secondary Outcome: Total Distance
Description: Subjects were instructed to walk on the treadmill and to tell the research coordinator to stop testing when they reached the point at which they typically would need to stop and sit down, or until 15 minutes had elapsed. When the subject reached their maximum distance, the treadmill testing was stopped. This was recorded as total distance based on number of minutes and seconds walked. Minutes was converted to meters based on calculation of defined speed of the treadmill.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: meters
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
meters | 237.49 (27.47) | 261.55 (27.47)

4. Secondary Outcome: Recovery Time
Description: After the subject completed the treadmill test they were asked to immediately return to the seated position. At this point a timer was started. When the subjects pain level returned to baseline (level of pain subject felt in a seated position before walking) the time was stopped. This was recorded as recovery time. Maximum recovery time is 15 minutes.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
minutes | 2.36 (.43) | 3.15 (.43)

5. Secondary Outcome: Area Under the Curve
Description: Subjects were instructed to walk on the treadmill and to tell the research coordinator to stop testing when they reached the point at which they typically would need to stop and sit down, or until 15 minutes had elapsed. At defined intervals (every 30 seconds) subjects were asked what their pain level was according to the NRS. The area under the curve of present pain intensity multiplied by the amount of time the subject walked.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale * minutes
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale * minutes | 100.59 (5.15) | 95.26 (5.15)

6. Secondary Outcome: Visual Analog Scale (VAS)
Description: The VAS asked subjects to place a mark indicative of their low back pain during the past day on a 100mm line, with 0mm representing no pain and 100mm representing extreme pain.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale | 52.31 (27.49) | 46.31 (24.44)

7. Secondary Outcome: Oswestry Disability Index (ODI) Score
Description: The ODI is a set of 10 questions each with five choices (maximum score of 5 points per question) designed to determine how back pain has affected the ability to manage everyday life (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and change positions). A total score range of 0-50; score of 0 indicates no disability and a score of 50 would indicate 100% disability.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale | 37.77 (2.76) | 36.49 (2.76)

8. Secondary Outcome: Swiss Spinal Stenosis (SSS) Score- Symptom Severity
Description: The SSS is a series of questions asking about symptom severity, physical function, and satisfaction. The symptom severity section is a set of 7 questions (maximum score is 5 points per question) and asks to rate pain for each question based on no pain, mild, moderate, severe or very severe pain. The total score (maximum=35) is added up and divided by seven. The maximum score for the symptom severity section (score=5) indicates very severe symptom severity.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale | 3.09 (.12) | 2.94 (.12)

9. Secondary Outcome: Swiss Spinal Stenosis- Physical Function
Description: The SSS is a series of questions asking about symptom severity, physical function, and satisfaction. The physical function section is a series of 5 questions (maximum 4 points per question) and asks to rate function for each question based on comfortably, sometimes with pain, always with pain, no functional ability. The total score (max=20) is divided by five. The maximum score for the physical function section (max=4) indicates no ability to function.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale | 2.40 (0.09) | 2.94 (0.09)

10. Secondary Outcome: Modified Brief Pain Inventory (mBPI)- Interference Score
Description: The mBPI is a series of questions that rates the severity and impact of pain on daily function. The questionnaire is made up of 4 pain severity items using the NRS scale, and seven pain interference sub-scales. The final interference score is an average of the seven sub-scales (0 indicating no interference and 10 indicating complete interference).
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale | 3.70 (0.42) | 3.58 (0.42)

11. Secondary Outcome: Roland Morris Disability Questionnaire
Description: The RMDQ consists of 24 yes/no statements about activity limitations due to back pain. These questions center on movement, ambulation, and self-care activities. Positive (yes) answers each contribute 1 point to cumulative score with total scores ranging from 0 (no disability) to 24 (severely disabled).
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale | 12.98 (.92) | 11.48 (.92)

12. Secondary Outcome: Patient Global Assessment (PGA)
Description: Subjects were asked to rate their low back pain according to the PGA. PGA is the impact of disease activity. PGA was measured on a 5-point scale, where 1=very good, 2=good, 3=fair, 4=poor, and 5=very poor.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Diphenhydramine
Number analyzed (Participants) | 26 | 26
units on a scale | 2.75 (.19) | 2.83 (0.19)

ADVERSE EVENTS:
Arm/Group | Pregabalin | Diphenhydramine
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 15/26 | 6/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=26) | Diphenhydramine (N=26)
Dizziness (General disorders) | 9 (9) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Somnolence (General disorders) | 5 (5) | 2 (2)
Dry mouth (General disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Peripheral edema (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No